CLINICAL TRIAL: NCT01242865
Title: Self Help Intervention to Decrease Stress: A Pilot Trial
Brief Title: Self Help Intervention to Decrease Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-006367
Record Dates: First submitted 2010-11-11; First posted 2010-11-17 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Stress, Psychological
Keywords: Stress; Anxiety; Resilience; Mindfulness; Quality of Life; Stress Management
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Attention and Interpretation Therapy (Other)
  Interventions: Behavioral: Attention and Interpretation Therapy

INTERVENTIONS:
Behavioral: Attention and Interpretation Therapy — Participants will receive a copy of the book, "Train Your Brain Engage Your Heart Transform Your Life" along with three handouts summarizing the contents of the book.
  Other Names: AIT; Stress Management Program

SUMMARY:
The present study is designed to test the feasibility and efficacy of a stand alone self help program for decreasing stress and anxiety and enhancing quality of life. The intervention will be offered in the form of a self help book and three handouts with no in-person instructor time.

DETAILED DESCRIPTION:
Stress is a ubiquitous problem and a mediator of symptoms for a variety of medical conditions. Most medical diagnoses, procedures, and physician visits are associated with considerable stress. Excessive stress is associated with adverse medical outcomes, unhealthy coping mechanisms, symptoms of anxiety and depression, and overall a poor quality of life. No specific pharmacologic treatment is available for treating stress. Further, it is often difficult or sometimes impossible to change the reality of circumstances causing stress in an individual. Thus increasing individual coping mechanisms and ability of a person to handle stress, rather than changing the stressors itself might be a more feasible approach towards reducing stress.

Several interventions are available to decrease stress. Majority of these programs entail extensive in-person training which impacts on widespread dissemination of the program. We are interested in applying an innovative approach toward stress management by testing the efficacy of a stand alone self help program offered in the form of a book with no in-person instructor time. Participants will receive a copy of the book, "Train Your Brain Engage Your Heart Transform Your Life" along with three handouts summarizing the contents of the book. This book describes the program of Attention and Interpretation therapy that is designed to help decrease stress and anxiety and has been developed at Mayo Clinic Rochester.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age
* Good general health
* Provided with, understand, and have signed the informed consent

Exclusion criteria:

* Are currently using (at time of enrollment) antipsychotics and/or antidepressants
* Have a life time history of schizophrenia.
* Previously participated in Attention and Interpretation Therapy (AIT) training.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of testing a self help stress management program for improving stress in a pilot clinical trial. | 12 Weeks

SECONDARY OUTCOMES:
To assess the efficacy of the self help stress management program on resilience. | 12 Weeks
To assess the efficacy of the self help stress management program on stress. | 12 Weeks
To assess the efficacy of the self help stress management program on anxiety. | 12 Weeks
To assess the efficacy of the self help stress management program on mindfulness. | 12 Weeks
To assess the efficacy of the self help stress management program on overall quality of life. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brent A. Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Sharma V, Bauer B, Prasad K, Sood A, Schroeder D. P02.197. Self help intervention to decrease stress and increase mindfulness: a pilot trial. BMC Complementary and Alternative Medicine 2012, 12(Suppl 1):P253. http://www.biomedcentral.com/1472-6882/12/S1/P253